CLINICAL TRIAL: NCT06479941
Title: Antibiotic Exposure During Pregnancy Affects Infant Gut Microbiota
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, xu xue, Vice Chief Physician, Peking University People's Hospital
Other Study IDs: PKUPH-X2
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Antibiotics Affecting Newborn Gut Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Umbilical cord blood, placenta, stool
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mother-infant cohort with antibiotic treatment group: E.g., Bacterial infection during pregnancy
  Interventions: Other: antibiotic treatment
- Mother-infant cohort (Prophylactic antibiotics therapy): E.g., cesarean section
  Interventions: Other: antibiotic treatment
- Mother-infant cohort (Natural delivery): E.g., Natural delivery
  Interventions: Other: antibiotic treatment

INTERVENTIONS:
Other: antibiotic treatment — AT: Mother-infant cohort with antibiotic treatment group CS: Mother-infant cohort (Prophylactic antibiotics therapy) ND: Mother-infant cohort (Natural delivery)

SUMMARY:
Based on a prospective birth cohort, the investigators will collect biological samples from participants including pregnant women and newborns, to measure the gut microbial diversity and metabolites of newborns. These results systematically evaluate the effects of antibiotic exposure on the structure and function of gut microbiota. The project can reveal the effects of antibiotic exposure on the growth and development of gut microbiota in early life.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant woman

   * aged 20-40 years old
   * natural conception
   * single pregnancy
   * gestational age ≥36 weeks
2. Newborn

   * normal Apgar score
   * no serious congenital diseases

Exclusion Criteria:

-

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pregnant woman registered in Peking University People's Hospital will plan to give birth in the hospital.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-06-25 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Infant gut microbiome | Pregnancy (12, 24, 37 weeks) and infants (born, 1 week, and 1, 3, 6, 12 months)
  * Diversity of gut microbiota
  * Abundance of antibiotic resistance genes in gut microbiota
  * Metabolic pathway of gut microbiota

SECONDARY OUTCOMES:
Antibiotic treatment | Pregnancy (12, 24, 37 weeks) and infants (born, 1 week, and 1, 3, 6, 12 months)
  * Frequency of antibiotic treatment
  * Kind and Dose of antibiotic;
  * Duration of antibiotic use;

CONTACTS AND LOCATIONS:
Locations (1):
- The Peking University People's Hospital, Beijing, China